CLINICAL TRIAL: NCT05317325
Title: A Translational Study of Tumor Antigen-pulsed Dendritic Cell Vaccine for Esophageal Squamous Cell Carcinoma
Brief Title: A Translational Study of Tumor Antigen-pulsed DC Vaccine for ESCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXDB-2203
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal cancer; tumour cell lysate; neoantigen; prime-boost; dendritic cell vaccine
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Autologous DCs pulsed with HOCl-oxidized autologous tumor lysate (OCDC) vaccine is administered in prime phase and personal neoantigen-sensitized DC(NeoDC) vaccine is administered in boost phase.
  Interventions: Biological: OCDC vaccine; NeoDC vaccine

INTERVENTIONS:
Biological: OCDC vaccine; NeoDC vaccine — OCDC vaccine and NeoDC vaccine are administered in a prime-boost regimen by subcutaneous injection.

SUMMARY:
The aim of this single center, single arm and prospective study is to explore the safety and efficacy of tumor antigen-pulsed DC vaccine( OCDC and NeoDC) for postoperative adjuvant treatment of ESCC

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of esophageal squamous cell carcinoma
* no preoperative adjuvant therapy
* Karnofsky performance status 0-2;
* The postoperative pathological stage is pT2-4 and / or N + M0 according to AJCC 8th
* Function of the main organs is normal;
* Edition Patient's written informed consent

Exclusion Criteria:

* Tumor emergencies;
* Abnormal coagulation function;
* Contagious diseases, such as HIV, HBV, HCV infection;
* Mental disorders;
* Concomitant tumors;
* Immunological co-morbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The number of treatment-related adverse events | From the first administration of vaccine to 3 months after the last administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Disease-free Survival | from the study start to 1 year after the study completion
  Number of participants with Disease-free Survival as assessed by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu Ding, Prof, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes